CLINICAL TRIAL: NCT00571389
Title: A Biospecimen Collection Study to Facilitate Development of an Ex-Vivo Device Platform for Culture, Immune Assay, and Biobanking of Leukapheresis-Derived Circulating Tumor Cells, Immune Cells, and Progenitor Cells.
Brief Title: A Biospecimen Collection Study of Leukapheresis-Derived Circulating Tumor Cells, Immune Cells, and Progenitor Cells.
Status: Recruiting | Type: Observational
Sponsor: BioCytics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BioCytics 0001; WIRB Protocol # 20070969
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor, Adult; Healthy Donors; COVID-19 Donors
Keywords: All Stages of cancer; All stages of solid tumor origin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral whole blood, immune cells, circulating tumor cells, discarded tissue obtained from biopsies and fluid (paracentesis, pleuracentesis), plasma-leukapheresis products, saliva, urine and stool.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Cancer Cohort: The first cohort of patients to be enrolled for this study will be adults (males and females) with histological proven solid tumors of any stage, seen for routine cancer care at participating community cancer clinic sites. Patients on clinical trials with experimental study drugs will be allowed to participate in this observational prospective study.
- Healthy Volunteer Cohort: Healthy volunteers make up the second, smaller study population for this observational biospecimen laboratory study. Healthy volunteers serve primarily to aid in the proficiency, quality control and/or optimization of study procedures, experimental design assay development, and for device/equipment validation.
- COVID-19 Disease Cohort: Due to the COVID-19 pandemic and the consequent amendment to aid in the research response, study subjects with COVID-19 disease may participate in all aspects of this protocol, but depending on their disease state, infection timeline, and age, participation may be limited to only one component, procedure, and/or type of biospecimen collection. Age is a very important criteria, as pediatric subjects (5-17 years old) will only be eligible to participate in minimally invasive biospecimen collection procedures.

SUMMARY:
Primary Objective:

This is a study to investigate the feasibility of harvesting, expanding, and selecting T lymphocytes from cancer patients and healthy volunteers. The preliminary objective of this study is aimed at selecting PD-1+ and CTLA4+ T cells and other cellular fractions from peripheral blood of cancer patients and healthy volunteers by using specific conjugated antibodies, evaluating their functional ex vivo anti-tumor cytotoxicity against targeted autologous tumor cells.

ELIGIBILITY:
Inclusion Criteria for Biospecimen(s) collection:

Cancer Cohort Inclusion Criteria:

1. Male or Female Adult ≥ 18 years of age.
2. Histological diagnosis of any solid tumor type and at any stage of disease progression including in the neoadjuvant/presurgical setting, adjuvant setting, or considered in remission.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 3 (see Appendix 2) and an estimated life expectancy of at least 3 months.
4. Subject or subject's legal representative provides written informed consent.
5. Negative serology screening test for HIV, Hepatitis B surface antigen, and Hepatitis C antibody, or negative reflex PCR test result for HIV, Hepatitis B Virus (HBV), and Hepatitis C Virus (HCV)
6. Additional eligibility criteria need to be met for leukapheresis collection:

   * ECOG Performance Status of 0 or 1 (see Appendix 2)
   * WBC ≥2000/μL
   * Neutrophils ≥1000/μL
   * Platelets ≥100x103/μL
   * Hemoglobin ≥9 g/dL
   * Creatinine ≤2.5 x ULN
   * AST ≤2.5 x ULN without, and ≤ 5 x ULN with hepatic metastases
   * Bilirubin ≤2 x ULN (except patients with Gilbert's syndrome, who must have total bilirubin ≤ 3.0 mg/dL)
   * Negative urine pregnancy test for women of childbearing potential

Healthy Volunteer Cohort Inclusion Criteria:

1. Male or Female Adult ≥ 18 years of age.

   ▪ Pediatric healthy volunteers from 5-17 years of age, with suspected or confirmed COVID-19 diagnosis by laboratory test will be eligible to participate in minimally invasive biospecimen collection procedures, as long as written parental consent has been obtained, and if applicable and technologically able, child assent. Minimally invasive biospecimen collection procedures allowed for pediatric participation include swabs (nasal, NP and OP), microcapillary sampling, and saliva or urine collection.
2. Healthy volunteers are eligible, including the following:

   * History of autoimmune disease or inflammatory disorder considered clinically stable by the Principal Investigator or treating physician's discretion.
   * Suspected or diagnosed COVID-19 disease by laboratory test, whether in the acute, sub-acute or convalesced state.
   * Employees of the study site(s) or BioCytics, as long as fulfilment of inclusion criteria 3.c is obtained.
3. Subject or subject's legal representative provides written informed consent.
4. Negative serology screening test for HIV, Hepatitis B surface antigen, and Hepatitis C antibody, or negative reflex PCR test result for HIV, HBV, and HCV.
5. Additional eligibility criteria need to be met for leukapheresis collection:

   * Must be ≥ 18 years of age.
   * WBC ≥2000/μL
   * Neutrophils ≥1000/μL
   * Platelets ≥100x103/μL
   * Hemoglobin ≥9 g/dL
   * Creatinine ≤2.5 x ULN
   * AST ≤2.5 x ULN
   * Bilirubin ≤2 x ULN (except patients with Gilbert's syndrome, who must have total bilirubin ≤ 3.0 mg/dL)
   * Negative urine pregnancy test for women of childbearing potential

2.3.4. Exclusion Criteria

1. Subjects with active infection requiring therapy (fever, localizing source) will be excluded until the infection resolves.

   a. This excludes subjects with suspected or confirmed COVID-19 by laboratory test while in the acute and sub-acute phase of viremia.
2. Underlying medical condition that, in the Principal Investigator's or treating oncologist's opinion, will obscure the interpretation of the patient's safety.
3. Confirmed positive reflex PCR test result for HIV, Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV).

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population of patients to be enrolled for this study will consist of two cohorts: 1) cancer patients, and to a lesser extent 2) healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2007-11; Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Carolina BioOncology Institute, Huntersville, North Carolina, United States

REFERENCES:
- See also: Related Info — http://www.carolinabiooncology.org

DOCUMENTS (1):
  • Study Protocol (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT00571389/Prot_000.pdf